CLINICAL TRIAL: NCT05371600
Title: The Effect of Preoperative Anxiolysis With Intravenous Midazolam on Intraoperative Sevoflurane Gas Consumption: A Prospective Randomized Controlled Study
Brief Title: Preoperative Anxiolysis With Intravenous Midazolam on Intraoperative Sevoflurane Gas Consumption
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ersel GULEC, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14949
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Midazolam; Sevoflurane
Keywords: Midazolam; Sevoflurane; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group M (Active Comparator): Patients receive midazolam IV at 0.04 mg/kg (group M).
  Interventions: Drug: Midazolam
- Group C (Placebo Comparator): Patients receive an equal volume of saline IV (group C, control group).
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Midazolam — midazolam IV at 0.04 mg/kg
  Arms: Group M
Other: Saline — an equal volume of saline IV
  Arms: Group C

SUMMARY:
This prospective, randomized, double-blind, placebo-controlled study is performed after obtaining written informed consent of patients who are scheduled for elective general surgery. After the admission to the preoperative unit 30 minutes before the surgery, The preoperative anxiety of patients is evaluated by The State-Trait Anxiety Inventory (STAI). Patients are randomly assigned to one of two groups in a 1:1 ratio by a computer-generated list. Patients receive midazolam IV at 0.04 mg/kg (group M) and an equal volume of saline IV (group C, control group). Anesthesia is induced with 2mg/kg of IV propofol. At a dose of 0.6 mg/kg, IV rocuronium bromide is given for neuromuscular blockade. Anesthesia is maintained at 2% sevoflurane. At the end of the surgery, anesthesia is terminated and the awake patients are extubated.

DETAILED DESCRIPTION:
An equal depth of anesthesia is achieved by evaluating an entropy value of 40-50 during the operation. Heart rate, blood pressure, the amount of sevoflurane consumed (ml), end-tidal sevoflurane concentration (%), sevoflurane MAC, inspiratory sevoflurane (%) are recorded at baseline and 15-minute intervals.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1 and 2
* patients who are scheduled for elective surgery
* BMI <30

Exclusion Criteria:

* history of psychiatric disease
* use of psychotropic medications
* neurological disorders
* cancer
* chronic pain
* cardiovascular, respiratory, and hepatic diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Sevoflurane consumption | 1 hour
  The amount of sevoflurane consumed (ml)

SECONDARY OUTCOMES:
end-tidal sevoflurane concentration (%) | 1 hour
  end-tidal sevoflurane concentration (%)

OTHER OUTCOMES:
sevoflurane MAC | 1 hour
  sevoflurane MAC
inspiratory sevoflurane (%) | 1 hour
  inspiratory sevoflurane (%)

CONTACTS AND LOCATIONS:
Overall Officials: Ersel Gulec, MD, Principal Investigator — Cukurova University
Locations (1):
- Department of Anesthesiology, Cukurova University Faculty of Medicine, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kil HK, Kim WO, Chung WY, Kim GH, Seo H, Hong JY. Preoperative anxiety and pain sensitivity are independent predictors of propofol and sevoflurane requirements in general anaesthesia. Br J Anaesth. 2012 Jan;108(1):119-25. doi: 10.1093/bja/aer305. Epub 2011 Nov 13. PMID 22084330
- [Background] Maranets I, Kain ZN. Preoperative anxiety and intraoperative anesthetic requirements. Anesth Analg. 1999 Dec;89(6):1346-51. doi: 10.1097/00000539-199912000-00003. PMID 10589606
- [Background] Melvin MA, Johnson BH, Quasha AL, Eger EI 3rd. Induction of anesthesia with midazolam decreases halothane MAC in humans. Anesthesiology. 1982 Sep;57(3):238-41. doi: 10.1097/00000542-198209000-00018. No abstract available. PMID 7114548
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167